CLINICAL TRIAL: NCT04330339
Title: Pilot Study to Assess Prolonged Nightly Fasting in Breast Cancer Survivors
Brief Title: Prolonged Nightly Fasting in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kully Family Foundation (Unknown)
Responsible Party: Principal Investigator, Elizabeth O'Donnell, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-586
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Fasting; Breast Cancer; Survivorship; Breast Cancer Recurrent
Keywords: Fasting; Breast Cancer; Survivorship; Breast Cancer Recurrent
MeSH Terms: conditions — Fasting; Breast Neoplasms | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental): * Eligible participants will undergo baseline assessments prior to starting the intervention.
    * Baseline assessments include measurements of weight, height, quality of life, fatigue, mood, levels of physical activity, and blood markers.
    * Participants will fast for 13 hours nightly for 12 weeks.
  * Assessments will be repeated at the completion of the 12-week intervention.
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — Fasting

SUMMARY:
This study is being done to examine whether fasting for 13 hours every night is feasible and if it can help breast cancer survivors lose weight and improve their health.

* Previous studies have found that women who are overweight or obese when their breast cancer is found (diagnosed) have a greater risk of their breast cancer recurring. Recent research suggests that prolonged nighttime fasting (>13 hours) may improve the risk of recurrence for breast cancer.
* This study will examine if fasting for 13 hours per night is doable for participants and will also study what the effect of fasting is on quality of life, mood, fatigue, body size, and markers of health in the blood.

DETAILED DESCRIPTION:
This research study involves fasting (not eating any food or drinking fluids that contain calories) for 13 hours nightly for 12 weeks.

* It is expected that about 40 people will take part in this research study.
* Eligible participants will undergo baseline assessments prior to starting the intervention.

  * Baseline assessments include measurements of weight, height, quality of life, fatigue, mood, levels of physical activity, and blood markers.
  * Assessments will be repeated at the completion of the 12-weeks

This is a a Feasibility Study, which means this is the first time that investigators are examining prolonged nightly fasting and its effect on breast cancer survivors body size, blood markers, quality of life, emotional regulation, fatigue and level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a documented history of histologically confirmed invasive breast cancer.
* Participants with a history of stage I to III invasive breast cancer, and no current evidence of disease.
* A history of bilateral breast cancer is allowed provided the patient is currently disease free, with stage I to III disease on both sides.
* No evidence of distant metastatic disease or unresectable locally recurrent disease
* All adjuvant or neoadjuvant cytotoxic chemotherapy, radiation, and surgery for breast cancer must have been completed at least 6 month prior to registration. Except:

  * Adjuvant hormonal therapy is permitted. Must have been on for a minimum of 1 month.
  * Adjuvant trastuzumab, pertuzumab, TDM1, or neratinib for Her2 positive breast cancer is permitted Age ≥18 years.
* Participant must be female.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Distant metastatic breast cancer (Stage IV breast cancer) or unresectable locally recurrent disease
* Participants with diabetes mellitus.
* Participants with a pre-existing eating disorder (anorexia nervosa, bulimia)
* Participants with a BMI< 19kg/m2 or a weight loss of 5% in the last month or 10% in the last 3 months.
* Participants using weight loss medications at the time of study enrollment.
* Participants using oral steroids at the time of enrollment.
* Participants who are receiving any other investigational agents. Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of prolonged fasting on the fetus are not known.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants adhere to 13 hours of fasting | 12 weeks
  Feasibility will be demonstrated if ≥60% of participants adhere to 13 hours of fasting nightly at least 70% of the nights during the intervention.
  Adherence will be assessed through patient-reported fasting logs.

SECONDARY OUTCOMES:
Change in body mass index (BMI) (kg/m^2) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (kg/m^2). Body mass index calculated using patient height (meters) and weight (kilograms) measured at baseline and at the completion of the study intervention. BMI = weight in kilograms divided by the square of height in meters.
Quality of life (QOL) Change using the Functional Assessment of Cancer Therapy General Scale (FACT-G) | 6 and 12 weeks
  FACT-G is a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences)
Change in Hospital Anxiety and Depression Scale (HADS) (min score: 0; max score: 21. A higher score indicates more anxiety and/or depression) | 6 and 12 weeks
  Effects of prolonged nightly fasting on psychological well-being using The Hospital Anxiety and Depression Scale (HADS). Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences)
Change in fatigue as assessed by Functional Assessment of Chronic Illness Therapy - Fatigue | 6 and 12 weeks
  13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. Higher scores represent better functioning or less fatigue.Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in physical activity using the Godin Leisure-Time Exercise Questionnaire | 6 and 12 weeks
  Calculated score where patient-reported weekly frequencies of strenuous, moderate, and light activities are multiplied by nine, five, and three, respectively. Total weekly leisure activity is calculated in arbitrary units by summing the products of the separate components, as shown in the following formula:
  Weekly leisure activity score = (9 x Strenuous) + (5 x Moderate) + (3 x Light)
Change in lipid profile | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences). (total cholesterol: mg/dL; triglycerides: mg/dL; high-density lipoprotein cholesterol mg/dL; low-density lipoprotein cholesterol mg/dL; very low-density lipoprotein cholesterol: mg/dL; cholesterol/HDL ratio mg/dL).
Change in hemoglobin A1c (%) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), hemoglobin A1c reported as percentage of average blood sugar level (mg/dL or mmol/L), higher % corresponds to higher average blood sugar levels (normal A1C level is below 5.7%)
Change in c-reactive protein (mg/L) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), mg/L (hs-CRP level of 1 mg/L or lower indicates low risk of CVD, hs-CRP level of 1-3 mg/L indicates moderate risk of CVD, hs-CRP level of greater than 3 mg/L indicates high risk of CVD)
Change in interleukin-6 (pg/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), pg/mL
Change in tumor necrosis factor alpha (pg/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), pg/mL
Change in insulin (mcU/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (mcU/mL)
Change in leptin (ng/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (ng/mL)
Change in adiponectin level (microgram/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (microgram/mL)
Change in insulin-like growth factor (ng/mL) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (ng/mL)
Change in homeostatic model assessment of insulin resistance (estimates beta cell function (%B) and insulin sensitivity (%S), as percentages of a normal reference population) | 12 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences). Plasma glucose: mmol/L (or mg/dL), Insulin: pmol/L (or microunits/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K O'Donnell, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Result] O'Donnell E, Shapiro Y, Comander A, Isakoff S, Moy B, Spring L, Wander S, Kuter I, Shin J, Specht M, Kournioti C, Hu B, Sullivan C, Winters L, Horick N, Peppercorn J. Pilot study to assess prolonged overnight fasting in breast cancer survivors (longfast). Breast Cancer Res Treat. 2022 Jun;193(3):579-587. doi: 10.1007/s10549-022-06594-4. Epub 2022 Apr 20. PMID 35441995